CLINICAL TRIAL: NCT01472081
Title: A Phase 1 Study of Nivolumab (BMS-936558) Plus Sunitinib, Pazopanib or Ipilimumab in Subjects With Metastatic Renal Cell Carcinoma
Brief Title: Nivolumab (BMS-936558; MDX-1106) in Combination With Sunitinib, Pazopanib, or Ipilimumab in Subjects With Metastatic Renal Cell Carcinoma (RCC) (CheckMate 016)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-016
Record Dates: First submitted 2011-10-26; First posted 2011-11-16 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Renal Cell Carcinoma; Clear-cell Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Clear-cell metastatic renal cell carcinoma | interventions — Nivolumab; pazopanib; Sunitinib; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm S: Nivolumab + Sunitinib (Experimental): Nivolumab 0.3, 2.0 (starting dose), 5.0 mg/kg solution intravenously every 21 days until Progressive disease (PD), toxicity or discontinue for other reasons
  Sunitinib 50 mg capsule by mouth on Days 1-28 of 42 day cycle until Progressive disease (PD), toxicity or discontinue for other reasons
  Interventions: Biological: Nivolumab; Drug: Sunitinib
- Arm P: Nivolumab + Pazopanib (Experimental): Nivolumab 0.3, 2.0 (starting dose), 5.0 mg/kg solution intravenously every 21 days until Progressive disease (PD), toxicity or discontinue for other reasons
  Pazopanib 800 mg tablet by mouth daily until Progressive disease (PD), toxicity or discontinue for other reasons
  Interventions: Biological: Nivolumab; Biological: Pazopanib
- Arm I-1: Nivolumab + Ipilimumab (Experimental): Nivolumab 3 mg/kg solution intravenously (IV) every 21 days during Induction phase and every 14 days during Maintenance phase until Progressive disease (PD), toxicity or discontinue for other reasons
  Ipilimumab 1mg/kg solution intravenously (IV) every 21 days during Induction phase (Ipilimumab will not be administered during Maintenance phase) until Progressive disease (PD), toxicity or discontinue for other reasons
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Arm I-3: Nivolumab + Ipilimumab (Experimental): Nivolumab 1mg/kg solution intravenously (IV) every 21 days during Induction phase and 3mg/kg solution intravenously (IV) every 14 days during Maintenance phase
  Ipilimumab 3mg/kg solution intravenously (IV) every 21 days during Induction phase. Ipilimumab will not be administered during Maintenance phase
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Arm IN-3: Nivolumab+Ipilimumab (Experimental): Nivolumab 3mg/kg solution intravenously (IV) every 21 days during Induction phase and 3mg/kg solution intravenously (IV) every 14 days during Maintenance phase
  Ipilimumab 3mg/kg solution intravenously (IV) every 21 days during Induction phase. Ipilimumab will not be administered during Maintenance phase
  Interventions: Biological: Nivolumab; Biological: Ipilimumab

INTERVENTIONS:
Biological: Nivolumab
  Other Names: BMS-936558 (MDX-1106)
Biological: Pazopanib
  Other Names: Votrient (Pazopanib hydrochloride)
  Arms: Arm P: Nivolumab + Pazopanib
Drug: Sunitinib
  Other Names: Sutent®; Sunitinib Malate
  Arms: Arm S: Nivolumab + Sunitinib
Biological: Ipilimumab
  Other Names: YERVOY™
  Arms: Arm I-1: Nivolumab + Ipilimumab; Arm I-3: Nivolumab + Ipilimumab; Arm IN-3: Nivolumab+Ipilimumab

SUMMARY:
The purpose is to determine the safety, effectiveness and best dose to use when giving Nivolumab in combination with Sunitinib, Pazopanib, or Ipilimumab for the treatment of metastatic renal cell carcinoma.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Subjects with histological confirmation of RCC
* Advanced or metastatic disease
* Measurable disease as defined by RECIST 1.1 criteria
* Karnofsky Performance Status (KPS) ≥80%
* Available tumor tissue (archival or recent acquisition)
* Subjects enrolled in the I-1, I-3 expansion arms and IN-3 addition arms must not have received any prior systemic therapy for RCC with the following exceptions:

  1. One prior adjuvant or neoadjuvant therapy for localized or locally advanced RCC is allowed provided recurrence occurred ≥ 6 months after the last dose of the adjuvant or neoadjuvant therapy
  2. Only prior cytokine based treatment for metastatic RCC [eg, interferon-alpha (IFN-alpha) or interleukin 2 (IL-2)] as prior therapy is allowed

Exclusion Criteria:

* Active central nervous system (CNS) metastases
* Active or history of autoimmune disease
* Ongoing symptomatic cardiac dysrhythmias or uncontrolled atrial fibrillation
* History of cerebrovascular accident including transient ischemic attack within the past 12 months
* History of pulmonary embolism or deep vein thrombosis (DVT) within the past 6 months
* Chronic systemic steroids (>10 mg/day Prednisone equivalents) or any other immunosuppressive agents
* White blood cell (WBC) <2,000/mm3
* Neutrophiles <1,500/mm3
* Platelets <100,000/mm3
* Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) >3x upper limit of normal (ULN)
* Total Bilirubin >1.5x ULN (except subjects with Gilbert syndrome, total bilirubin <3.0 mg/dL)
* Cardiac ejection fraction <LLN (lower limit of normal)
* Serum creatinine >1.5x ULN or creatinine clearance <40 mL/min (Cockroft-Gault formula)

Exclusion Criteria for Arm S and Arm P only:

* For dose escalation cohorts - subjects who received prior Sunitinib or Pazopanib and required permanent discontinuation due to toxicity or required dose reduction or delay during the first 12 weeks of therapy due to toxicity, or received both prior Sunitinib and Pazopanib
* Poorly controlled hypertension
* Active bleeding or bleeding susceptibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2012-02-09 (Actual); Primary Completion 2016-02-02 (Actual); Study Completion 2021-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- United States (10):
  - City Of Hope, Duarte, California
  - Sidney Kimmel Comprehensive Cancer Center At Johns Hopkins, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Nassau, New York, New York
  - Blumenthal Cancer Center, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - University Of Texas M.D. Anderson Cancer Center, Houston, Texas
- Canada (4):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario

REFERENCES:
- [Derived] Amin A, Plimack ER, Ernstoff MS, Lewis LD, Bauer TM, McDermott DF, Carducci M, Kollmannsberger C, Rini BI, Heng DYC, Knox J, Voss MH, Spratlin J, Berghorn E, Yang L, Hammers HJ. Safety and efficacy of nivolumab in combination with sunitinib or pazopanib in advanced or metastatic renal cell carcinoma: the CheckMate 016 study. J Immunother Cancer. 2018 Oct 22;6(1):109. doi: 10.1186/s40425-018-0420-0. PMID 30348216
- [Derived] Dorff TB, Pal SK, Quinn DI. Novel tyrosine kinase inhibitors for renal cell carcinoma. Expert Rev Clin Pharmacol. 2014 Jan;7(1):67-73. doi: 10.1586/17512433.2014.862496. Epub 2013 Dec 2. PMID 24308791
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 194 participants were enrolled; 153 were treated. Participants were enrolled but not treated due to the following reasons: withdrawal of consent (n=5), no longer met study criteria (n=32), administrative reason by sponsor (n=1), or other reasons (n=3)
Groups:
- Arm S: SUN + NIV2: Nivolumab 2 mg/kg administered on Day 1 and 22 of each 6 week (42 day) cycle as a 1-hour IV infusion followed 60 minutes later with Sunitinib 50 mg orally on Day 1 - 28 of each 42 day cycle until Progressive Disease (PD), toxicity or discontinuation for other reasons.
- Arm S: SUN + NIV5: Nivolumab 5 mg/kg administered on Day 1 and 22 of each 6 week (42 day) cycle as a 1-hour IV infusion followed 60 minutes later with Sunitinib 50 mg orally on Day 1 - 28 of each 42 day cycle until Progressive Disease (PD), toxicity or discontinuation for other reasons.
- Arm P: PAZ + NIV2: Nivolumab 2 mg/kg administered on Day 1 and 22 of each 6 week (42 day) cycle as a 1-hour IV infusion followed 60 minutes later with Pazopanib 800 mg orally on Day 1 - 42 of each 42 day cycle until Progressive Disease (PD), toxicity or discontinuation for other reasons.
- Arm I-1: IPI1 + NIV3: Induction: Nivolumab 3 mg/kg was administered as a 1-hour IV infusion followed by Ipilimumab 1 mg/kg administered IV infusion over 90 minutes every 3 weeks for 4 doses.
  Maintenance: Nivolumab 3 mg/kg was administered as a 1-hour IV infusion every 2 weeks, starting 3 weeks after the 4th dose of induction therapy or after Day 113 if the 4th dose of induction therapy had not been administered due to treatment delays.
- Arm I-3: IPI3 + NIV1: Induction: Nivolumab 1 mg/kg was administered as a 1-hour IV infusion followed by Ipilimumab 3 mg/kg administered IV infusion over 90 minutes every 3 weeks for 4 doses.
  Maintenance: Nivolumab 3 mg/kg was administered as a 1-hour IV infusion every 2 weeks, starting 3 weeks after the 4th dose of induction therapy or after Day 113 if the 4th dose of induction therapy had not been administered due to treatment delays.
- Arm IN-3: IPI3 + NIV3: Induction: Nivolumab 3 mg/kg was administered as a 1-hour IV infusion followed by Ipilimumab 3 mg/kg administered IV infusion over 90 minutes every 3 weeks for 4 doses.
  Maintenance: Nivolumab 3 mg/kg was administered as a 1-hour IV infusion every 2 weeks, starting 3 weeks after the 4th dose of induction therapy or after Day 113 if the 4th dose of induction therapy had not been administered due to treatment delays.
Period: Overall Study
Arm/Group | Arm S: SUN + NIV2 | Arm S: SUN + NIV5 | Arm P: PAZ + NIV2 | Arm I-1: IPI1 + NIV3 | Arm I-3: IPI3 + NIV1 | Arm IN-3: IPI3 + NIV3
Started | 7 | 26 | 20 | 47 | 47 | 6
Completed | 0 | 0 | 0 | 1 | 0 | 0
Not Completed | 7 | 26 | 20 | 46 | 47 | 6
Not completed — Continuing treatment at time of analysis | 1 | 4 | 1 | 8 | 9 | 0
Not completed — Disease Progression | 4 | 10 | 12 | 31 | 22 | 3
Not completed — Study drug toxicity | 2 | 9 | 4 | 6 | 13 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event unrelated to study drug | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Poor/non-compliance | 0 | 0 | 1 | 0 | 1 | 0
Not completed — No longer meets study criteria | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Subject request to discontinue treatment | 0 | 3 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm S: SUN + NIV2 | Arm S: SUN + NIV5 | Arm P: PAZ + NIV2 | Arm I-1: IPI1 + NIV3 | Arm I-3: IPI3 + NIV1 | Arm IN-3: IPI3 + NIV3 | Total
Number analyzed (Participants) | 7 | 26 | 20 | 47 | 47 | 6 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (11.36) | 58.3 (8.62) | 56.3 (8.52) | 53.0 (8.97) | 55.6 (11.58) | 54.8 (2.71) | 55.4 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 7 | 2 | 14 | 9 | 1 | 33
  Male | 7 | 19 | 18 | 33 | 38 | 5 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 1 | 2 | 1 | 6
  Not Hispanic or Latino | 7 | 22 | 18 | 42 | 40 | 5 | 134
  Unknown or Not Reported | 0 | 2 | 2 | 4 | 5 | 0 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 2 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 1 | 1 | 0 | 5
  White | 6 | 22 | 18 | 44 | 45 | 6 | 141
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With AEs, SAEs, and AEs Leading to Discontinuation
Description: Safety assessments by treatment arm and dose level were based on incidence of AEs, and the incidence of serious adverse events (SAEs). AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4= Potentially Life-threatening or disabling.
Time Frame: From date of first dose to date of last dose plus 100 days (assessed up to March 2016, approximately 49 months)
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Arm S: SUN + NIV2 | Arm S: SUN + NIV5 | Arm P: PAZ + NIV2 | Arm I-1: IPI1 + NIV3 | Arm I-3: IPI3 + NIV1 | Arm IN-3: IPI3 + NIV3
Number analyzed (Participants) | 7 | 26 | 20 | 47 | 47 | 6
participants
  All-causality SAEs (any grade) | 3 | 16 | 13 | 29 | 30 | 4
  All-causality SAEs (grade 3-4) | 1 | 14 | 10 | 20 | 24 | 4
  Drug-related SAEs (any grade) | 2 | 12 | 2 | 11 | 16 | 3
  Drug-related SAEs (grade 3-4) | 0 | 10 | 2 | 9 | 16 | 3
  All-cause AEs led to discontinuation (any grade) | 3 | 10 | 5 | 5 | 15 | 2
  All-cause AEs led to discontinuation (grade 3-4) | 2 | 9 | 4 | 3 | 11 | 0
  All-Causality AEs (any grade) | 7 | 26 | 20 | 47 | 47 | 6
  All-Causality AEs (grade 3-4) | 6 | 24 | 16 | 33 | 34 | 6
  Drug-related AEs (any grade) | 7 | 26 | 20 | 43 | 45 | 6
  Drug-related AEs (grade 3-4) | 5 | 22 | 14 | 18 | 29 | 5

2. Secondary Outcome: Best Overall Response Rate (BOR)
Description: BOR was defined as the best response designation over the study as a whole, recorded between the date of first dose of study medication and the date of objectively documented progression per RECIST 1.1 criteria or the date of subsequent anti-cancer therapy, whichever occurred first.
  CR = Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm. PR = At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD = At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression. SD = Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: From date of first dose to date of disease progression or subsequent anti-cancer therapy, whichever occurred first (assessed up to March 2016, approximately 49 months)
Population: All treated participants
Measure: Number; unit: percentage of participants
Arm/Group | Arm S: SUN + NIV2 | Arm S: SUN + NIV5 | Arm P: PAZ + NIV2 | Arm I-1: IPI1 + NIV3 | Arm I-3: IPI3 + NIV1 | Arm IN-3: IPI3 + NIV3
Number analyzed (Participants) | 7 | 26 | 20 | 47 | 47 | 6
percentage of participants
  Complete Response | 1 | 0 | 1 | 5 | 0 | 0
  Partial Response | 5 | 11 | 8 | 14 | 19 | 0
  Stable Disease | 1 | 11 | 7 | 19 | 17 | 5
  Progressive Disease | 0 | 1 | 4 | 8 | 8 | 1
  Unable to Determine | 0 | 3 | 0 | 1 | 3 | 0

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the proportion of participants who achieved a BOR of either complete response (CR) or partial response (PR) in the population of interest.
  CR = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR = At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of first dose to interim analysis (Assessed up to March 2016, approximately 49 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm S: SUN + NIV2 | Arm S: SUN + NIV5 | Arm P: PAZ + NIV2 | Arm I-1: IPI1 + NIV3 | Arm I-3: IPI3 + NIV1 | Arm IN-3: IPI3 + NIV3
Number analyzed (Participants) | 7 | 26 | 20 | 47 | 47 | 6
percentage of participants | 85.7 [42.1 to 99.6] | 42.3 [23.4 to 63.1] | 45.0 [23.1 to 68.5] | 40.4 [26.4 to 55.7] | 40.4 [26.4 to 55.7] | 0 [0 to 0]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was computed for participants with BOR of CR or PR only, and defined as the time between the date of first documented objective response and the date of the first subsequent disease progression or death. Participants who remained alive and had not progressed were censored on the last tumor assessment date (prior to subsequent cancer therapy).
Time Frame: From date of first dose to date of disease progression or death, whichever occurred first (assessed up to March 2016, approximately 49 months)
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Arm S: SUN + NIV2 | Arm S: SUN + NIV5 | Arm P: PAZ + NIV2 | Arm I-1: IPI1 + NIV3 | Arm I-3: IPI3 + NIV1 | Arm IN-3: IPI3 + NIV3
Number analyzed (Participants) | 7 | 26 | 20 | 47 | 47 | 6
weeks | 45.6 [18.14 to NA] — Upper 95% CI not reached | 78.1 [36.14 to NA] — Upper 95% CI not reached | 30.1 [12.14 to 174.14] | 88.7 [37.14 to NA] — Upper 95% CI not reached | 85.9 [35.14 to NA] — Upper 95% CI not reached | NA [NA to NA] — No participants in this arm achieved BOR of PR or CR

5. Secondary Outcome: Rate of Progression-free Survival (PFS) at Week 24
Description: Rate of PFS at week 24 was defined as the proportion of participants remaining progression free or surviving at 24 weeks, calculated by the product-limit method (Kaplan-Meier estimate) which took into account censored data. Participants who did not have any on-study tumor assessment and did not die were censored on the date of first dose of study medication.
Time Frame: 24 weeks
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants with PFS
Arm/Group | Arm S: SUN + NIV2 | Arm S: SUN + NIV5 | Arm P: PAZ + NIV2 | Arm I-1: IPI1 + NIV3 | Arm I-3: IPI3 + NIV1 | Arm IN-3: IPI3 + NIV3
Number analyzed (Participants) | 7 | 26 | 20 | 47 | 47 | 6
Percentage of participants with PFS | 100 [100 to 100] | 72.9 [49.3 to 86.8] | 54.9 [29.4 to 74.6] | 55.6 [40.0 to 68.6] | 63.8 [48.4 to 75.7] | NA [NA to NA] — PFS rate at 24 weeks was not calculated for this arm

6. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of first dose of study medication to the date of first disease progression or death. Participants who did not have any on-study tumor assessment and did not die were censored on the date of first dose of study medication.
Time Frame: as for outcome 4
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm S: SUN + NIV2 | Arm S: SUN + NIV5 | Arm P: PAZ + NIV2 | Arm I-1: IPI1 + NIV3 | Arm I-3: IPI3 + NIV1 | Arm IN-3: IPI3 + NIV3
Number analyzed (Participants) | 7 | 26 | 20 | 47 | 47 | 6
months | 11.3 [7.62 to NA] — Upper 95% CI not reached | 12.7 [5.55 to 19.38] | 7.2 [2.79 to 11.07] | 7.7 [3.71 to 14.29] | 9.4 [5.62 to 18.63] | 8.5 [1.31 to NA] — Upper 95% CI not reached

ADVERSE EVENTS:
Time Frame: From first dose to date of last dose plus 100 days
Groups:
- SUNITINIB+NIVOLUMAB: Nivolumab (2mg/kg or 5mg/kg)administered on Day 1 and 22 of each 6 week (42 day) cycle as a 1-hour IV infusion followed 60 minutes later with Sunitinib 50 mg orally on Day 1 - 28 of each 42 day cycle until Progressive Disease (PD), toxicity or discontinuation for other reasons.
- PAZOPANIB+NIVOLUMAB: Nivolumab 2 mg/kg administered on Day 1 and 22 of each 6 week (42 day) cycle as a 1-hour IV infusion followed 60 minutes later with Pazopanib 800 mg orally on Day 1 - 42 of each 42 day cycle until Progressive Disease (PD), toxicity or discontinuation for other reasons.
- NIVO 3+IPI 1 (MG/KG): Induction: Nivolumab 3 mg/kg was administered as a 1-hour IV infusion followed by Ipilimumab 1 mg/kg administered IV infusion over 90 minutes every 3 weeks for 4 doses.
  Maintenance: Nivolumab 3 mg/kg was administered as a 1-hour IV infusion every 2 weeks, starting 3 weeks after the 4th dose of induction therapy or after Day 113 if the 4th dose of induction therapy had not been administered due to treatment delays.
- NIVO 1+IPI 3 (MG/KG): Induction: Nivolumab 1 mg/kg was administered as a 1-hour IV infusion followed by Ipilimumab 3 mg/kg administered IV infusion over 90 minutes every 3 weeks for 4 doses.
  Maintenance: Nivolumab 3 mg/kg was administered as a 1-hour IV infusion every 2 weeks, starting 3 weeks after the 4th dose of induction therapy or after Day 113 if the 4th dose of induction therapy had not been administered due to treatment delays.
- NIVO 3+IPI 3 (MG/KG): Induction: Nivolumab 3 mg/kg was administered as a 1-hour IV infusion followed by Ipilimumab 3 mg/kg administered IV infusion over 90 minutes every 3 weeks for 4 doses.
  Maintenance: Nivolumab 3 mg/kg was administered as a 1-hour IV infusion every 2 weeks, starting 3 weeks after the 4th dose of induction therapy or after Day 113 if the 4th dose of induction therapy had not been administered due to treatment delays.
Arm/Group | SUNITINIB+NIVOLUMAB | PAZOPANIB+NIVOLUMAB | NIVO 3+IPI 1 (MG/KG) | NIVO 1+IPI 3 (MG/KG) | NIVO 3+IPI 3 (MG/KG)
Serious Adverse Events (participants affected / at risk) | 19/33 | 13/20 | 29/47 | 30/47 | 4/6
Other Adverse Events (participants affected / at risk) | 33/33 | 20/20 | 47/47 | 46/47 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SUNITINIB+NIVOLUMAB (N=33) | PAZOPANIB+NIVOLUMAB (N=20) | NIVO 3+IPI 1 (MG/KG) (N=47) | NIVO 1+IPI 3 (MG/KG) (N=47) | NIVO 3+IPI 3 (MG/KG) (N=6)
Methaemoglobinaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Hypopituitarism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0
Autoimmune colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 6 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 4 | 6 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Erosive duodenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0
Hernia (General disorders) | 1 | 0 | 0 | 0 | 0
Mucosal ulceration (General disorders) | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 4 | 0
Pyrexia (General disorders) | 1 | 2 | 4 | 3 | 2
Sudden death (General disorders) | 0 | 1 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1 | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 2 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2 | 1 | 1 | 0
Pneumonia legionella (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 4 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 4 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 2 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 2 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 1 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 0 | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 6 | 2 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0 | 1 | 1
Transient global amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 0 | 3 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SUNITINIB+NIVOLUMAB (N=33) | PAZOPANIB+NIVOLUMAB (N=20) | NIVO 3+IPI 1 (MG/KG) (N=47) | NIVO 1+IPI 3 (MG/KG) (N=47) | NIVO 3+IPI 3 (MG/KG) (N=6)
Anaemia (Blood and lymphatic system disorders) | 8 | 3 | 7 | 10 | 1
Leukopenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 5 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0 | 2 | 2 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 2 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 2 | 2 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 1 | 6 | 3 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 5 | 2 | 1
Ear congestion (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 2 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 2 | 6 | 2
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 1 | 1
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Endocrine disorder (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 5 | 0 | 3 | 8 | 3
Hypothyroidism (Endocrine disorders) | 10 | 4 | 10 | 13 | 5
Lymphocytic hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 2 | 0 | 0 | 2 | 0
Eye pain (Eye disorders) | 0 | 1 | 1 | 0 | 1
Lacrimation increased (Eye disorders) | 4 | 0 | 3 | 5 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0 | 1 | 2 | 1
Periorbital oedema (Eye disorders) | 5 | 0 | 1 | 1 | 0
Photopsia (Eye disorders) | 0 | 2 | 2 | 1 | 0
Vision blurred (Eye disorders) | 2 | 1 | 6 | 5 | 1
Visual impairment (Eye disorders) | 1 | 1 | 1 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 2 | 2 | 2 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 4 | 4 | 5 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 7 | 10 | 12 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 4 | 3 | 1
Anal inflammation (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Autoimmune colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Breath odour (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 1
Constipation (Gastrointestinal disorders) | 9 | 8 | 14 | 14 | 2
Defaecation urgency (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 21 | 14 | 12 | 25 | 5
Dry mouth (Gastrointestinal disorders) | 11 | 2 | 5 | 8 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 11 | 5 | 6 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 2 | 3 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 6 | 1 | 5 | 3 | 2
Gastritis (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 | 3 | 4 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 4 | 0 | 0 | 2 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 2 | 3 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 20 | 16 | 19 | 26 | 4
Oral pain (Gastrointestinal disorders) | 5 | 4 | 1 | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 8 | 2 | 7 | 0 | 2
Toothache (Gastrointestinal disorders) | 2 | 2 | 3 | 2 | 0
Vomiting (Gastrointestinal disorders) | 10 | 9 | 15 | 14 | 3
Asthenia (General disorders) | 0 | 1 | 3 | 4 | 1
Chest discomfort (General disorders) | 3 | 2 | 2 | 2 | 0
Chest pain (General disorders) | 0 | 3 | 5 | 1 | 1
Chills (General disorders) | 8 | 6 | 13 | 9 | 3
Face oedema (General disorders) | 4 | 0 | 1 | 1 | 1
Fatigue (General disorders) | 29 | 15 | 31 | 35 | 6
Generalised oedema (General disorders) | 2 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 3 | 0 | 2 | 2 | 0
Localised oedema (General disorders) | 1 | 1 | 0 | 1 | 0
Malaise (General disorders) | 2 | 2 | 1 | 1 | 1
Mucosal inflammation (General disorders) | 11 | 5 | 2 | 4 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 2 | 0 | 1
Oedema (General disorders) | 1 | 1 | 2 | 1 | 1
Oedema peripheral (General disorders) | 11 | 5 | 12 | 13 | 3
Pain (General disorders) | 0 | 2 | 2 | 2 | 1
Pyrexia (General disorders) | 10 | 7 | 18 | 11 | 6
Sensation of foreign body (General disorders) | 2 | 0 | 0 | 0 | 0
Temperature intolerance (General disorders) | 2 | 1 | 2 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 2 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infected bite (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 2 | 1 | 1 | 2 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 4 | 3 | 0
Skin infection (Infections and infestations) | 1 | 1 | 1 | 1 | 0
Tinea infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 3 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 7 | 9 | 7 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 2 | 3 | 2
Vulvitis (Infections and infestations) | 0 | 0 | 2 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 5 | 0 | 2 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 5 | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 1 | 3 | 3 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 13 | 5 | 8 | 16 | 3
Amylase increased (Investigations) | 5 | 0 | 4 | 8 | 2
Aspartate aminotransferase increased (Investigations) | 12 | 6 | 9 | 14 | 3
Blood alkaline phosphatase increased (Investigations) | 5 | 3 | 2 | 4 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 2 | 3 | 1
Blood cholesterol increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 12 | 2 | 7 | 9 | 2
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 2 | 0 | 11 | 19 | 2
Lymphocyte count decreased (Investigations) | 9 | 1 | 1 | 4 | 1
Neutrophil count decreased (Investigations) | 6 | 0 | 1 | 1 | 0
Platelet count decreased (Investigations) | 6 | 0 | 3 | 0 | 0
Weight decreased (Investigations) | 4 | 4 | 5 | 11 | 4
Weight increased (Investigations) | 3 | 0 | 7 | 4 | 1
White blood cell count decreased (Investigations) | 7 | 1 | 1 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 16 | 11 | 13 | 19 | 5
Dehydration (Metabolism and nutrition disorders) | 7 | 6 | 7 | 9 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 4 | 5 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 4 | 7 | 8 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 2 | 5 | 4 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 5 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 2 | 1 | 4 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 5 | 3 | 6 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 9 | 1 | 6 | 6 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 2 | 3 | 6 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 9 | 24 | 12 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 6 | 15 | 8 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 8 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2 | 1
Lower extremity mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 5 | 3 | 4 | 3
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 6 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 6 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 3 | 5 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 5 | 11 | 10 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 8 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 6 | 8 | 5 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1 | 0
Ataxia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Cerebellar syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 3 | 1
Disturbance in attention (Nervous system disorders) | 2 | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 11 | 3 | 10 | 12 | 2
Dysgeusia (Nervous system disorders) | 21 | 10 | 5 | 8 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 13 | 5 | 15 | 13 | 4
Hyperaesthesia (Nervous system disorders) | 1 | 2 | 0 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 4 | 2 | 1 | 3 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 4 | 3 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 0 | 3 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 3 | 1
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 2 | 0
Speech disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 2 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 3 | 2 | 2
Anxiety (Psychiatric disorders) | 3 | 2 | 7 | 4 | 1
Confusional state (Psychiatric disorders) | 2 | 0 | 2 | 1 | 0
Depression (Psychiatric disorders) | 4 | 0 | 1 | 2 | 2
Insomnia (Psychiatric disorders) | 5 | 4 | 9 | 9 | 3
Irritability (Psychiatric disorders) | 1 | 1 | 0 | 3 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 2 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 1 | 1 | 2 | 1
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 2 | 1 | 2 | 1
Nocturia (Renal and urinary disorders) | 0 | 1 | 1 | 3 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 2 | 1 | 2 | 0
Polyuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 4 | 1 | 3 | 6 | 2
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 13 | 24 | 14 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 7 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 4 | 13 | 9 | 2
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 7 | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 9 | 6 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 6 | 5 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 5 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 8 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 2 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 7 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 3 | 11 | 4 | 1
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 2 | 2 | 4 | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 6 | 4 | 1 | 0 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 5 | 2 | 3
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 4 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 13 | 0 | 1 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 9 | 18 | 21 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 9 | 7 | 18 | 15 | 4
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 | 4 | 7 | 8 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 4 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 1 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 2 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 0 | 0
Yellow skin (Skin and subcutaneous tissue disorders) | 7 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 5 | 3 | 3 | 6 | 1
Haematoma (Vascular disorders) | 1 | 1 | 0 | 1 | 0
Hot flush (Vascular disorders) | 5 | 2 | 3 | 4 | 0
Hypertension (Vascular disorders) | 17 | 8 | 4 | 6 | 3
Hypotension (Vascular disorders) | 2 | 4 | 3 | 6 | 2
Orthostatic hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Autoimmune hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Genital infection fungal (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Libido decreased (Psychiatric disorders) | 2 | 0 | 0 | 2 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.